CLINICAL TRIAL: NCT02754609
Title: Hookworm Therapy for Coeliac Disease: A Phase 1B Safety and Dose-ranging Clinical Trial Examining Sustained Gluten Consumption in Hookworm-naive and Hookworm-infection People With Coeliac Disease
Brief Title: Hookworm Therapy for Coeliac Disease
Acronym: NainCeD-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Cook University, Queensland, Australia (Other)
Collaborators: Townsville Hospital (Other Government); The Prince Charles Hospital (Other Government); Christchurch Hospital (Other); Logan Hospital, Queensland (Other Government); Australian Institute of Tropical Health and Medicine (Other); QIMR Berghofer Medical Research Institute (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-2016-CTN-01363-1
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Necator americanus; Helminths; Autoimmunity; Clinical Trials, Phase I; Randomized Controlled Trial
MeSH Terms: conditions — Celiac Disease; Autoimmune Diseases | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Placebo, 20 hookworm L3 or 40 hookworm L3
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Re-identifiable IP containers
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Necator americanus-hookworm larvae L3-10 (Experimental): A total of 40 participants week 0 and week 8 will have low dose hookworms present in 2-3 drops of water applied to their skin and then covered in a light dressing. The hookworms are Necator americanus-hookworm larvae L3; 10 L3 in 200 microliter (uL) of deionized water presented in an Eppendorf tube. All participants will undergo interventions of Gluten free diet, Gluten micro-challenge, Inadvertent gluten challenge and Moderate gluten challenge. At week 42, participants will have the option of going on the liberal diet.
  Interventions: Other: Gluten micro-challenge; Other: Inadvertent gluten challenge; Other: Moderate gluten challenge; Other: Liberal diet; Other: Necator americanus-hookworm larvae L3-10; Other: Gluten free diet
- Tabasco® Sauce (Placebo Comparator): A total of 10 participants at week 0 and week 8 will have Tabasco® Sauce present in 2-3 drops of water applied to their skin and covered in a light dressing. Tabasco® Sauce is an ideal placebo as the sensation to the skin is similar to a hookworm. All participants will undergo interventions of Gluten free diet, Gluten micro-challenge, Inadvertent gluten challenge and Moderate gluten challenge.
  Interventions: Other: Gluten micro-challenge; Other: Inadvertent gluten challenge; Other: Moderate gluten challenge; Other: Tabasco® Sauce; Other: Gluten free diet
- Necator americanus-hookworm larvae L3-20 (Experimental): A total of 10 participants at week 0 and week 8 will have medium dose hookworms present in 2-3 drops of water applied to their skin and then covered in a light dressing. The hookworms are Necator americanus-hookworm larvae L3; 20 L3 in 200 uL of deionized water presented in an Eppendorf tube. All participants will undergo interventions of Gluten free diet, Gluten micro-challenge, Inadvertent gluten challenge and Moderate gluten challenge. At week 42, participants will have the option of going on the liberal diet.
  Interventions: Other: Gluten micro-challenge; Other: Inadvertent gluten challenge; Other: Moderate gluten challenge; Other: Liberal diet; Other: Necator americanus-hookworm larvae L3-20; Other: Gluten free diet

INTERVENTIONS:
Other: Gluten micro-challenge — From week 12 to week 24, all participants will start a gluten micro-challenge from 10mg/day for the first 2 weeks escalating over the this period to 50mg/day at the end of week 24.
Other: Inadvertent gluten challenge — From week 24 to week 36, all participants will be on gluten 50mg/day and 1g twice weekly.
Other: Moderate gluten challenge — From week 36 to week 42, all participants will be on gluten 2g/day.
Other: Liberal diet — From week 42, all participants will be unblinded and those who have received hookworm therapy have the option to go on a liberal diet of more than 10g of gluten/day from week 42 to week 94.
  Arms: Necator americanus-hookworm larvae L3-10; Necator americanus-hookworm larvae L3-20
Other: Necator americanus-hookworm larvae L3-10 — A total of 40 participants at week 0 and week 8 will have hookworms L3-10 present in 2-3 drops of water applied to their skin and then covered in a light dressing.
  Arms: Necator americanus-hookworm larvae L3-10
Other: Tabasco® Sauce — Arm: Placebo Comparator: Tabasco® Sauce A total of 10 participants at week 0 and week 8 will have Tabasco® Sauce present in 2-3 drops of water applied to their skin and covered in a light dressing
  Arms: Tabasco® Sauce
Other: Necator americanus-hookworm larvae L3-20 — A total of 40 participants at week 0 and week 8 will have hookworms L3-20 present in 2-3 drops of water applied to their skin and then covered in a light dressing.
  Arms: Necator americanus-hookworm larvae L3-20
Other: Gluten free diet — From week 0 to week 12, all participants will be on a gluten free diet.

SUMMARY:
This trial is a Phase 1b multicentre, multinational, randomized, double-blind with single-blind arm and open label extension phase, placebo controlled, clinical trial evaluating the safety and predictability of an escalating gluten consumption to activate Coeliac Disease (CeD) in (a) a small cohort of people with diet-managed CeD treated with a placebo (n=10), and in (b) cohorts following low (L3-10; n=40) and medium (L3-20; n=10) dose hookworm inocula.

The investigators 4 aims for the study are:

Aim 1: Undertake a multiple-phase and escalating gluten challenge assessing safety to gluten exposure in hookworm-naïve and hookworm-infected people with CeD.

Aim 2: This phase Ib study recognizes that the evidence supporting this novel intervention is rudimentary and addresses amongst others the following questions: (a) The importance of L3 dose on Participant health, and (b) the importance of L3 dose on the safety of escalating gluten challenge and (c) the need for a comparator group should a phase II trial be warranted.

Aim 3: Examine the changes in intestinal T cell responses induced by hookworm infection and gluten exposure.

Aim 4: Assess the impact of hookworm infection and purified hookworm-derived proteins on gluten peptide-specific immune responses ex vivo.

DETAILED DESCRIPTION:
This trial is a Phase 1b multicentre, multinational, randomized, double-blind with single-blind arm and open label extension phase, placebo controlled, clinical trial evaluating the safety and predictability of an escalating gluten consumption to activate Coeliac Disease (CeD) in (a) a small cohort of people with diet-managed CeD treated with a placebo (n=10), and in (b) cohorts following low (L3-10; n=40) and medium (L3-20; n=10) dose hookworm inocula.

Aim 1&2/Clinical study: The primary outcome will be the safety of an escalating 30-week gluten challenge in hookworm naïve or hookworm infected people with CeD following a medium-high dose hookworm infection, assessed by the change of duodenal villous height to crypt depth ratio (V:C) between pre-trial (week -2) and post-challenge (week 42). This will be a binary variable defined as safe if gluten challenge is completed and V:C ratio >2.0 and there is <20% change in its value from baseline or fail if drop out occurs prior to the completion of the gluten challenge or V:C ratio is <2.0 or its change from baseline is >20%.

Secondary outcomes include safety of low and medium intensity hookworm infection at intermediate (12 weeks and 24 weeks) endpoints of an escalating gluten challenge, assessed by incidence of adverse events, serious adverse events as well as general health. Secondary outcome measures include changes in V:C ratio from baseline to intermediate endpoints, progression through successful gluten challenge phases of the trial including a liberal diet, mucosal intraepithelial lymphocyte count, Celiac Symptom Index (CSI questionnaire), Celiac-Quality of Life Score (QOL questionnaire) and the serum immunoglobulin A (IgA) tissue transglutaminase (tTG) level of all cohorts.

Aims 3&4/Associated in vitro cell measures and ex vivo mucosal stimulation investigations: The associated studies are designed to more fully explore the immunological processes underpinning the clinical outcomes, and to take advantage of mucosal tissue collected in excess of the clinical requirements to test individual components of hookworm secretions which we believe hold great potential as future therapies. These experiments are complex and often depend on the quality of tissue and the cells collected.

Study Procedure: After written informed consent is obtained at the screening visit and prior to enrolment Participants may require some haematological work to confirm eligibility. Participants will be randomized to receive hookworm larvae (L3-10 or L3-20) suspended in 2-3 drops of water applied to the skin and covered with a light dressing, or Tabasco® Sauce in solution (Placebo Comparator). Before inoculation, each Participant will complete a QOL questionnaire, submit a fresh faecal specimen, and undergo a blood draw and duodenal biopsy. Thereafter each week for the duration of participation, a food diary and CSI questionnaire will be submitted. At designated times, gluten will be introduced in escalating volumes. Blood, faecal and biopsy collections, and a QOL questionnaire will also be collected. To better evaluate the independent effect of L3 on host immunity, the L3-20 cohort will undergo an endoscopy at week 12 in lieu of the week 36 intervention.

Safety Parameters/Analysis: General health assessments, physical examination and vital signs will be obtained at screening and thereafter at designated clinic visits (or symptom driven as required). Incidence and severity of Adverse and Serious Events including evidence of gluten intolerance and hookworm related complications of Participants will be evaluated formally through structured questionnaires (CSI weekly and QOL at the designated times) to be scrutinised by the designated research nurse and informally through Participant initiated personal contact with a research nurse or clinician. As well, blood for clinical safety and histological results will be scrutinised contemporaneously (by a designated research nurse or designated researcher) for incidence and severity of laboratory abnormalities. Blood results and symptom scores will be coded in a re-identifiable format before adding to an access-restricted and secure database. Screening blood tests to include serum pregnancy test at screening (a positive test will exclude the Participant from entering the trial) and urine pregnancy test if pregnancy is suspected throughout the trial. The 12-month progression to a liberal diet will be monitored by tTG evaluated monthly, with monthly CSI evaluation and Participant contact.

Laboratory Parameters/Analysis: Blood analysis: Complete blood count (CBC), IgA-tTG titre, liver and renal function and iron tests and a screening serum pregnancy test will be performed at Sullivan Nicolaides Pathology (SNP) in Australia and Canterbury Health Laboratories in New Zealand. From the residual blood, peripheral blood mononuclear cells will be harvested (when circumstances permit) and serum will be stored.

Faecal analysis: Samples will be collected in anaerobic collection bags with an aliquot to be transferred into a provided screw top plastic jar, both to be frozen at -20°C for short term storage and transport, and stored at -80°C long-term for parasite egg quantitative polymerase chain reaction (qPCR) analysis to be performed by nominated un-blinded personnel supervised by Prof. James McCarthy at QIMR Berghofer Medical Research Institute, with the results to remain blinded to all other trial personnel. Faecal samples will also be stored for future analysis of bacterial communities (the microbiota).

Mucosal analysis: Duodenal biopsies (14 pinch biopsies, consistent with previous trials) will be taken by a nationally and trial accredited gastroenterologist supported by a sedationist in an accredited facility. Four biopsies will be committed for conventional histology. To ensure standardisation the Biopsy forceps to be used will be Boston Scientific Radial Jaw® 4 - 2.8mm. Paraffin embedded tissue sections (3 μm) will be stained with H&E and anti-cluster of differentiation 3 (anti-CD3). Clinical histopathology will be supervised by a specialist in gastrointestinal pathology (A/Prof. Andrew Clouston) and reported contemporaneously for clinical purposes. Best representative field images from each case will be selected by Prof. Clouston, then coded in re-identifiable format before adding to an access-restricted and secure database, and later scored for intraepithelial lymphocytes (IEL)% and V:C by a single pathologist (Dr. Greg Miller). At each time point, two four biopsy tissue samples will be stored at -80°C in 10% glycerolRNA stabilisation solution for future gene expression and microbiota analyses.

Total Blood volume: 50 ml per collection x 6 from week minus 4 to week 42. 10 ml per month for 12 months. Total 420 ml over 2 years.

Sample size determination: Gluten consumption is toxic when consumed by people with CeD. Unlike a conventional trial testing an intervention to reverse disease, this trial relies on gluten toxicity to promote disease activity. The trial primarily evaluates the safety of gluten exposure in CeD in hookworm-infected Participants. The escalating gluten challenge proposed is unprecedented, and whilst liberal gluten consumption is consumed by many people with CeD either though ignorance of diagnosis or a conscious decision not to comply with medical advice, it is anticipated this challenge will adversely affect the unprotected placebo controls. Consistent with this concern, the control cohort has been kept small. The study will consist of 60 participants, with 10 in the control group, 40 in the low-dose hookworm group (L3-10) and 10 in the medium-dose hookworm group (L3-20).

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent and is willing to comply with all Protocol scheduled visits, treatment plan, laboratory tests, and other trial procedures and in the opinion of the Investigator has a good understanding of the Protocol, the length of the study and the demands of the study.
2. Aged between 18-80 (at time of consent);
3. Have a pre-treatment histological diagnosis of Marsh grade 3 CeD;
4. Have a pre-trial V:C >2.0;
5. Have elevated tTG or endomysial Ab +ve pre-trial;
6. Have been adherent to a gluten-free diet for >6 months pre-enrolment;
7. Have a tTG <20 IU/mL (normal <15) at screening;
8. Have a CSI <35 at screening;
9. If female, has met either of criterion "a or b" below:

   1. If of non-childbearing potential, has met 1 of the following - Amenorrheic for at least 2 years, or has had a hysterectomy and/or bilateral oophorectomy at least 8 weeks prior to screening, or has had a tubal ligation at least 8 weeks prior to screening.
   2. If of childbearing potential, must be willing to use the acceptable methods of contraception and abide by the timelines as indicated
10. In the opinion of the Investigator is in good general health

Exclusion Criteria:

1. Have any finding at screening that in the opinion of the Investigator or medical monitor would compromise the safety of the Participant or affect their ability to adhere to protocol scheduled visits, treatment plan, laboratory tests, and other trial procedures.
2. Have participated in any other clinical trial and/or have received an investigational drug or device within 30 days of screening.
3. Have history or current evidence of any of the following: compromised respiratory function (chronic obstructive pulmonary disease, respiratory depression, signs or symptoms of hypoxia at screening); thyroid pathology (unless stabilized and euthyroid for >3 months at the time of screening); hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection; evidence of clinically significant chronic cardiac, hepatic or renal disease; psychiatric illness (poorly controlled); seizure disorder or any other chronic health issues that in the opinion of the Investigator would exclude the Participant from the trial.
4. History of substance abuse or current substance abuse that in the opinion of the Investigator would exclude the Participant from the trial.
5. Have a history of intolerance, allergy or hypersensitivity to the proposed placebo - Tabasco® Sauce or any of its known ingredients.
6. Have a history of intolerance, allergy or hypersensitivity to the proposed anthelmintic - mebendazole.
7. Have a history of intolerance, allergy or hypersensitivity to the proposed chemicals used in preparation of N.americanus - amphotericin B and Betadine that in the opinion of the Investigator would exclude the Participant from the trial.
8. Current requirement for consistent use of anti-inflammatory drugs (includes prescription and over the counter medication >2 doses per week, that in the opinion of the Investigator would significantly alter the Participant's immunity), aspirin exceeding 125 mg/day or the use of immunotherapeutics;
9. Diagnosis of cancer which has been in remission for < 5 years, excluding Participants with adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
10. Poor venous access making the Participant unable to comply with the safety laboratory testing and/or endoscopy sedation requirements.
11. Are an employee of the Sponsor, Investigator or study centre or immediate family of such employees or the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Safety of 30-week gluten challenge | 44 weeks
  The primary outcome will be the safety of an escalating 30-week gluten challenge in hookworm naïve or hookworm infected people with CeD following a medium-high dose hookworm infection, assessed by the change of duodenal villous height to crypt depth ratio (V:C) between pre-trial (week -2) and post-challenge (week 42). This will be a binary variable defined as safe if gluten challenge is completed and V:C ratio >2.0 and there is <20% change in its value from baseline or fail if drop out occurs prior to the completion of the gluten challenge or V:C ratio is <2.0 or its change from baseline is >20%.

SECONDARY OUTCOMES:
Difference in mucosal intraepithelial lymphocyte count between baseline (week -2) and week 42 | 14 weeks
  This secondary outcome is the mucosal intraepithelial lymphocyte count measured from tissue collected per-endoscopy comparing baseline (week -2) to week 42 to assess the safety of administrating hookworms vs placebo.
Difference in V:C ratio between baseline (week -2) and week 42 | 14 weeks
  This secondary outcome assesses the duodenal mucosal villous height to crypt depth ratio (V:C) measured from tissue collected per-endoscopy comparing baseline (week -2) to week 42 to assess the safety of administrating hookworms vs placebo.
Difference in mucosal intraepithelial lymphocyte count between baseline (week -2) and week 42 | 38 weeks
  This secondary outcome is the mucosal intraepithelial lymphocyte count measured from tissue collected per-endoscopy comparing baseline (week -2) to week 42 to assess the effect of medium level of gluten exposure in participants who have received placebo or L3-10 hookworms.
Difference in mucosal intraepithelial lymphocyte count between baseline (week -2) and week 36 | 44 weeks
  This secondary outcome is the mucosal intraepithelial lymphocyte count measured from tissue collected per-endoscopy comparing baseline (week -2) to week 36 to assess the effect of intermittent gluten in all participants.
Difference in mucosal intraepithelial lymphocyte count between baseline (week -2) and week 94 | 96 weeks
  This secondary outcome is the mucosal intraepithelial lymphocyte count measured from tissue collected per-endoscopy comparing baseline (week -2) to week 94 to assess the effect of a liberal diet in participants who have received hookworm L3-10 or L3-20 hookworms.
Difference in Celiac Symptom Index (CSI Questionnaire) between baseline (week 0) and week 36 | 36 weeks
  This secondary outcome is the analysis of the weekly CSI questionnaire from baseline (week 0) to week 36 to assess the effect of inadvertent gluten in all participants.
Difference in Celiac Symptom Index (CSI Questionnaire) between baseline (week 0) and week 42 | 42 weeks
  This secondary outcome is the analysis of the weekly CSI questionnaire from baseline (week 0) to week 42 to assess the effect of moderate gluten in all participants.
Difference in Celiac Symptom Index (CSI Questionnaire) between baseline (week 0) and week 94 | 94 weeks
  This secondary outcome is the analysis of the weekly CSI questionnaire from baseline (week 0) to week 42 to assess the effect of a liberal diet in participants who have received L3-10 or L3-20 hookworms.
Difference in Celiac-Quality of Life Score (QOL questionnaire) between baseline (week 0) and week 36 | 36 weeks
  This secondary outcome is the analysis of the QOL questionnaire from baseline (week 0) to week 36 to assess the effect of inadvertent gluten in all participants.
Difference in Celiac-Quality of Life Score (QOL questionnaire) between baseline (week 0) and week 42 | 42 weeks
  This secondary outcome is the analysis of the QOL questionnaire from baseline (week 0) to week 42 to assess the effect of moderate gluten in all participants.
Difference in Celiac-Quality of Life Score (QOL questionnaire) between baseline (week 0) and week 94 | 94 weeks
  This secondary outcome is the analysis of the QOL questionnaire from baseline (week 0) to week 94 to assess the effect of a liberal diet in participants who have received L3-10 or L3-20 hookworms.
Difference in Immunoglobulin A tissue transaminase (tTG) between baseline (week -4) and week 36 | 40 weeks
  This secondary outcome is the analysis of the Immunoglobulin A tissue transaminase (tTG) level measured in serum from baseline (week -4) to week 36 to assess the effect of inadvertent gluten in all participants.
Difference in Immunoglobulin A tissue transaminase (tTG) between baseline (week -4) and week 42 | 46 weeks
  This secondary outcome is the analysis of the Immunoglobulin A tissue transaminase (tTG) level measured in serum from baseline (week -4) to week 42 to assess the effect of moderate gluten in all participants.
Difference in Immunoglobulin A tissue transaminase (tTG) between baseline (week -4) and week 94 | 98 weeks
  The secondary outcome is the analysis of the Immunoglobulin A tissue transaminase (tTG) level measured in serum from baseline (week -4) to week 94 to assess the effect of a liberal diet in participants who have received L3-10 or L3-20 hookworms.
Difference in V:C ratio between baseline (week -2) and week 24 | 38 weeks
  This secondary outcome assesses the duodenal mucosal villous height to crypt depth ratio (V:C) measured from tissue collected per-endoscopy comparing baseline (week -2) to week 24 to assess the effect of trace gluten in participants who have received placebo or L3-10 hookworms.
Difference in V:C ratio between baseline (week -2) and week 94 | 96 weeks
  This secondary outcome assesses the duodenal mucosal villous height to crypt depth ratio (V:C) measured from tissue collected per-endoscopy comparing baseline (week -2) to week 94 to assess the effect of a liberal diet in participants who have received L3-10 or L3-20 hookworms.
Difference in V:C ratio between baseline (week -2) and week 12 | 14 weeks
  This secondary outcome assesses the duodenal mucosal villous height to crypt depth ratio (V:C) measured from tissue collected per-endoscopy comparing baseline (week -2) to week 12 to assess the safety of administrating L3-20 hookworms.

CONTACTS AND LOCATIONS:
Overall Officials: John Croese, MBBS, MD, Principal Investigator — Prince Charles Hospital
Locations (4):
- Australia (3):
  - Prince Charles Hospital, Brisbane, Queensland
  - Logan Hospital, Logan City, Queensland
  - Townsville Hospital, Townsville, Queensland
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No